CLINICAL TRIAL: NCT00291109
Title: Quantitative Real Time PCR in Cytolytic Formalin Fixed Breast Cells Obtained by Periareolar Fine Needle Aspiration. An Ancillary Protocol to a Chemoprevention Trial of Letrozole
Brief Title: An Examination of Predictors of Indicators of Response to Letrozole 2.5 mg
Status: Completed | Type: Observational
Sponsor: University of Kansas (Other)
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 9298
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Breast Cancer
Keywords: breast atypia; breast epithelial hyperplasia; Ki-67; RTPCR; microdissection
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: letrozole 2.5 mg

SUMMARY:
To assess the quantitative real time PCR results of oligonucleotide probes for a number of gene transcription products that may be useful as predictors or indicators of response to letrozole

DETAILED DESCRIPTION:
To assess the quantitative real time PCR results of oligonucleotide probes for a number of gene transcription products (PCNA, cyclin-D1, ER alpha, PR, pS2, 450 aromatase, bcl-2, bax, caspase-3, and VEGFR) that may be useful as predictors or indicators of response to letrozole

ELIGIBILITY:
Inclusion Criteria:

* evidence of hyperplasia with/without atypia upon random periareolar fine needle aspiration of breast
* on hormone replacement therapy
* postmenopausal
* increased risk of developing breast cancer based on personal or family history
* never have taken aromatase inhibitors or selective estrogen receptor modulators in last six months
* women who have a high risk of breast cancer
* older than 18 years

Exclusion Criteria:

* no anticoagulants
* no marked breast tenderness
* not pregnant or within twelve months of breast feeding/childbirth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-01; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States